CLINICAL TRIAL: NCT05225974
Title: A Phase 1 Study of Liraglutide Injection and Victoza® in Healthy Chinese Subjects: An Open, Randomized, Single-Dose and Crossover Study
Brief Title: A Randomized Phase 1 Study of Liralutide Injection in Healthy Chinese Subjects
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: The Affiliated Hospital of Qingdao University (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Crossover | Masking: None | Purpose: Other
Other Study IDs: NBT-1698-P1
Record Dates: First submitted 2022-01-28; First posted 2022-02-07 (Actual); Last update posted 2022-02-07 (Actual); Status verified 2022-01

CONDITIONS: Therapeutic Equivalency
Keywords: Liraglutide;Pharmacokinetic;bioequivalence
MeSH Terms: interventions — Liraglutide

STUDY DESIGN:
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Liraglutide injection (Experimental)
  Interventions: Drug: Liraglutide injection
- Liraglutide injection(Victoza®) (Active Comparator)
  Interventions: Drug: Liraglutide injection(Victoza®)

INTERVENTIONS:
Drug: Liraglutide injection — At a single dose of 0.6 mg of Liraglutide injection by subcutaneous injection
  Arms: Liraglutide injection
Drug: Liraglutide injection(Victoza®) — At a single dose of 0.6 mg of Liraglutide injection(Victoza®) by subcutaneous injection
  Arms: Liraglutide injection(Victoza®)

SUMMARY:
The study was designed as a single-site, randomized, open-label, crossover under fasted conditions. A single oral dose of 0.6 mg Liraglutide injection and Victoza® was given to the 32 healthy Chinese adult male volunteers.Blood samples were collected up to 72 h after administration.The primary pharmacokinetic endpoints were AUC0-t, AUC0-∞, and Cmax. Safety profile and immunogenicity data were collected from each subject.

DETAILED DESCRIPTION:
The study was designed as a single-site, randomized, open-label, crossover under fasted conditions. A single oral dose of 0.6 mg Liraglutide injection and Victoza® was given to the 32 healthy Chinese adult male volunteers.Volunteers were randomized 1:1 at the beginning to receive a single 0.6 mg dose of Victoza® or Liraglutide injection by subcutaneous injection during the first period. Following 7 days washout period, all subjects received the alternate formulation during the second period. Blood samples were collected up to 72 h after administration.The primary pharmacokinetic endpoints were AUC0-t, AUC0-∞, and Cmax. Safety profile and immunogenicity data were collected from each subject.

ELIGIBILITY:
Inclusion Criteria:

* Healthy male vulunteers aged 18 and above.
* The body mass index is in the range of 19.0-26.0 kg/m2 (including the critical value).
* Before the study, all subjects have been informed of the study's purpose, protocal, benefits, and risks, and signed the informed consent voluntarily.

Exclusion Criteria:

* Medical examinations revealed clinically significant abnormalities or any evidence or history of clinically significant disease.
* Volunteers who had used systemic glucocorticoid drugs within 3 months before enrollment.
* Participation in another clinical trial within 3 months.
* Smoking more than 5 cigarettes per day during the 3 months prior to screening.
* Blood donation, massive blood loss (#400mL) or enrolled in other clinical trials 3 months prior to screening.
* Any use of other prescription drugs (including contraceptive)#over-thecounter drugs, Chinese herbal medicine, health care products and 30 days prior to medication for this study.

Min Age: 18 Years | Sex: Male | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 32 (Actual)
Dates: Start 2021-07-16 (Actual); Primary Completion 2021-07-30 (Actual); Study Completion 2021-08-19 (Actual)

PRIMARY OUTCOMES:
Peak Plasma Concentration (Cmax) | 40 days
  Evaluation of Peak Plasma Concentration (Cmax)
Area under the plasma concentration versus time curve (AUC)0-t | 40 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-t
Area under the plasma concentration versus time curve (AUC)0-∞ | 40 days
  Evaluation of Area under the plasma concentration versus time curve (AUC)0-∞

SECONDARY OUTCOMES:
Incidence of Treatment-Emergent Adverse Events | 40 days
  Collection of adverse events

CONTACTS AND LOCATIONS:
Locations (1):
- Phase I Clinical Research Center, Qingdao, Shandong, China